CLINICAL TRIAL: NCT03696498
Title: Effects of PArtial Excavation in One Procedure Versus Partial Excavation in Two Procedures of PRImary Deep CAries in Permanent Teeth - A Randomised, Multicenter Clinical Superiority Trial With Blinded Outcome Assessment
Brief Title: Effects of Partical Excavation in One Versus Two Procedures of Primary Deep Caries (PAPRICA)
Acronym: PAPRICA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Public Dental Health Care System, Denmark (Other); Malmö University, Sweden (Unknown); Halmstad County Hospital (Other); Karolinska Institutet (Other); Göteborg University (Other); Lithuania (Unknown)
Responsible Party: Principal Investigator, Lars Bjørndal, Associate professor, PhD, dr odont, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: THE PAPRICA TRIAL
Record Dates: First submitted 2017-05-08; First posted 2018-10-04 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Primary Dental Caries
Keywords: Partial excavation; Deep dentin caries; RCT

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Partial caries excavation (1 step) (Experimental): Patients with radiographical caries within the pulpal ¼ of the dentine with the presence of a radiodense zone separating the pulp from the demineralised dentine is candidates for the treatment. Local anaesthesia shall be used. as this procedure is identical for the two interventions tested in this trial. A partial removal of carious dentine is performed with superficial removal of the outermost infected and necrotic part of the demineralised dentine.
  Intervention: A permanent resin restoration is placed on top of the remained caries.
  Interventions: Procedure: Resin restoration (1 step)
- Partial caries excavation (2 steps) (Active Comparator): Patients with radiographical caries within the pulpal ¼ of the dentine with the presence of a radiodense zone separating the pulp from the demineralised dentine is candidates for the treatment. Before randomisation, the participants receive the first excavation procedure as this procedure is identical for the two interventions tested in this trial. A partial removal of carious dentine is performed with superficial removal of the outermost infected and necrotic part of the demineralised dentine.
  Intervention: After randomisation, a calcium hydroxide containing base material is used and a temporary glass-ionomer restoration is placed in the entire cavity. After 4-6 months, the temporary restoration is removed, final excavation is carried out with hand excavators until firm but stained dentine remains, and a permanent resin restoration is placed.
  Interventions: Procedure: Resin restoration (2 steps)

INTERVENTIONS:
Procedure: Resin restoration (1 step) — Permanent resin restoration is placed on top of the partial removed caries.
  Arms: Partial caries excavation (1 step)
Procedure: Resin restoration (2 steps) — A calcium hydroxide containing base material is used and a temporary glass-ionomer restoration is placed in the entire cavity. After 4-6 months the patients are recalled. The temporary restoration is removed and final excavation is carried out with hand excavators until firm but stained dentine remains. A permanent resin restoration is performed.
  Arms: Partial caries excavation (2 steps)

SUMMARY:
Background: Deep caries is the most frequent reason for performing root canal treatments. Minimally invasive methods for the treatment of deep carious lesions might therefore be relevant to avoid pulp exposures and consequently to prevent root canal treatments. A 2 step carious removal approach has shown to avoid exposures. But we do not know whether a selective removal of carious tissue in well-defined deep caries lesions involving the pulpal quarter of the dentin can be successfully completed in 1 step.

Objectives: To investigate partial (selective) excavation by 1 vs 2 step in the treatment of deep caries in permanent teeth.

Design: RCT multinational superiority study with 2 parallel groups and blinded outcome assessment. The allocation sequence for partial (selective) carious removal vs 2 step stepwise carious removal (1:1) will be centralized and computer-generated, stratified for age and centre and concealed for the investigators.

Inclusion criteria: children (≥9 years) and adults with primary well-defined deep caries in a permanent tooth. The lesion should reach the pulpal ¼ of the dentin with presence of a radiodense zone on a bitewing.

Exclusion criteria: spontaneous and prolonged pain within the last 6 months; pain causing disturbed night sleep; negative pulp test; apical radiolucency; restoration in close contact with pulp; the patient has communication problems; no written informed consent.

Experimental intervention: 1-step selective carious removal to soft or firm dentine at central site , and peripheral non selective carious removal to hard dentin followed by a permanent resin restoration. Control intervention: Stepwise excavation (2- step, involving first step which is identical to the experimental intervention but a base material and a temporary glass-ionomer restoration is placed. The amount removed is as much as a proper restoration can be placed. After 4-6 months the patients are recalled and the temporary restoration is removed and final selective carious removal is completed until firm dentin remains followed by permanent resin restoration.

The primary outcome is to avoid pulp complication at the 1-year follow-up evaluating. The secondary outcomes are to arrest caries progression and sufficient restoration at the 1-year follow-up. All outcomes will further be assessed 3 years after inclusion.

DETAILED DESCRIPTION:
Originality of the project: The originality of the PAPRICA project will be to provide high-quality clinical evidence for optimal treatment of deep caries lesions which is urgently needed. The project is very relevant within an area that has been known for suggestions of many treatments with the most invasive ones being the most popular ones. Only few previous studies define the depth of the carious lesion, data on well-defined lesions will clarify guidelines. Also, our design of this trial will attempt to reduce the risk of bias which is always critical when the investigator can't be blinded. In this respect the randomization will first be initiated after the 1 step of carious removal is completed. Results from a systematic review and a recent meta-analysis support stepwise excavation compared to complete excavation. However, firm evidence for one visit selective caries removal to soft dentine (previously defined as partial excavation) is still lacking. The project will for the first time investigate the caries treatment dilemma within a broader clinical context and thus aiming to reduce number of dental visits and to reduce acute pain. In the PAPRICA project a well-defined selective caries removal to soft dentine will be used as the lack of definitions are frequent in previously published clinical trials.

With this study we are aiming to 1) improve the treatment of deep caries by markedly reducing tooth-related pain, and consequently reduce the number of sick days due to toot-related pain; 2) reduce the number, complexity and duration of dental visits needed to treat deep caries; 3) provide data for an updated evidence-based treatment guideline for an improved health-care system.

Selection of participants: All patients at a participating clinical trial site are considered for participation. Patients will be eligible, if they comply with well-defined inclusion and exclusion criteria.

Statistical plan and data analysis: Sample size is 668 patients, based on the primary outcome 'pulp complications' among controls being 25%, and 15% in the experimental group, and combined with a type-I error of 5%; and a type-II error of 10%. Blinded interim analyses will be carried out. Statistical analysis of data from outcome measures - the gained frequencies of treatments leading to preservation of vital tooth without pain, apical pathology and no root filling will be examined using logistic regression analysis to assess the treatment effect adjusted for stratification variables. Odds ratio estimates will be used with 95% CI. Missing data will be handled using multiple imputations.

Randomization: Only one deep caries lesion per patient will be randomized. The trial will use block randomization with the following to stratifications variables: 1) Center; 2) Age (9-20 years/over 20 years). The randomization in the PAPRICA trial will be performed using an online system.

Blinding: The investigator performing the follow-up examination is not the same who performed the treatment. The analysis of the radiographs of the tooth at follow-up is carried out by an observer-committee being blinded for the intervention. The statistical analyses are carried out blinded. Patient blinding is not possible as the two intervention groups are performed as either a one-treatment procedure or a two-treatment procedure.

The patients who will be randomly allocated to 1-step partial caries removal will receive a treatment that normally is not practiced in relation to deep caries. However, there is a lack of randomised clinical trials investigating, whether partial caries removal has a positive prolonged effect with respect to maintained vital pulp and absence of apical pathology. The possible gain with the proposed treatment concept could be that the treatment of deep caries could be rationally performed without an extra treatment session and it may to a larger extent lead to an avoidance of exposure to the pulp. Patients who will be randomly allocated to 2-step partial caries removal receive a well-known treatment of deep caries. The intention is that we will gain data to reduce the risk of pulp exposures and thus the number of root canal treatments and possible reduce the number of days 'out-of' work due to tooth pain following an unnecessary invasive treatment of deep caries

Discontinuation and withdrawal: If a patient does not show-up for an appointment, attempts to make a re-appointment are carried out up to 3 times. It is important to stress that great effort should be carried out in order to find reasons for not attending an established appointment or if a patient wishes to withdraw from the trial. he investigators shall discontinue a participant from the trial intervention at any time, if: 1) There are signs of caries progression or failure of the restoration; 2) The participant is diagnosed with any of the exclusion criteria during the intervention period (except 'deep carious tooth has restoration in close contact with pulp'); 3) The participant experiences intolerable adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children >9 years.
* Primary coronal caries without pain in a permanent tooth (pain is accepted when evoked by a hot, cold, or sweet stimulus of short duration and disappears when the stimulus is removed).
* The radiograph shows caries within the pulpal ¼ of the dentine with the presence of a radiodense zone separating the pulp from the demineralised dentine.
* No exposure of the pulp following the first excavation.
* Available for recall at 1 and 3 years.
* Written informed consent.

Exclusion Criteria:

* Actual deep carious tooth presenting spontaneous and/or prolonged pain within the last 6 months, or pain causing disturbed night sleep.
* Actual deep carious tooth with negative thermal and/or electrical pulp test.
* Radiograph shows apical or radicular radiolucency of the tooth.
* Deep carious tooth has restoration in close contact with pulp.
* No written informed consent.

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2015-01; Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pulp complications | 3 years
  Pulp complications will be assessed using a registration scheme: no pulp vitality, based on negative thermal and/or electric pulp test; apical radiolucency as assessed by the blinded examiner based on radiograph; pulp exposure due to treatment of signs of pulpitis; endodontic treatment (root filling).
Restoration quality | 3 years
  Quality of restorations will be assessed using af registration scheme: intact restoration: Intact restoration, Total lost of restoration; Partly Lost of restoration

CONTACTS AND LOCATIONS:
Overall Officials: Lars Bjørndal, Dr odont, PhD, Study Director — University of Copenhagen
Locations (11):
- Denmark (8):
  - PDHS - Bornholm, Rønne, Bornholm
  - PDHS - Gentofte, Gentofte Municipality, Charlottenlund
  - University of Copenhagen, Copenhagen, Copenhagen N
  - PDHS - Copenhagen municipality, Copenhagen, Copenhagen V
  - PDHS - Randers municipality, Randers, Randers C
  - PDHS - Hørsholm, Hørsholm, Rungsted Kyst
  - PDHS - Aarhus municipality, Aarhus, Viby J
  - PDHS - Brøndby, Brøndby
- University of Norway - Lithuania, Klaipėda, Lithuania
- Preventive Dentistry Department, Moscow, Dolgorukovskaya, Russia
- Malmo University, Malmo, Malmo C, Sweden

IPD SHARING:
Plan to Share IPD: Yes